CLINICAL TRIAL: NCT05071846
Title: An Open Label, Single Arm, Phase I Clinical Study Assessing Safety, Tolerability, and Efficacy of MVX-ONCO-2 in Patients With Advanced Solid Tumors
Brief Title: MVX-ONCO-2 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Eugenio Fernandez, Dr Med, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVX-2021-01
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MVX-ONCO-2 (Experimental): Implantation of 2 capsules containing MVX-2 cells and 1 injection of 4 × 10^6 lethally irradiated autologous tumor cells
  Interventions: Biological: MVX-ONCO-2

INTERVENTIONS:
Biological: MVX-ONCO-2 — One administration of MVX-ONCO-2 (or vaccination) consists of the implantation of 2 capsules containing MVX-2 cells and 1 injection of 4 × 10^6 lethally irradiated autologous tumor cells. Tumor cells will have prealably been harvested from the participant through a surgical procedure.
  A full treatment course with MVX-ONCO-2 consists of a total of 6 vaccinations: 4 vaccinations 1 week apart, followed by 2 boosters 2 weeks apart. Capsules are removed 1 week after implantation.

SUMMARY:
MVX-ONCO-2 is a patient-specific, cell-based, active immunotherapy where the participant's immune response to their own tumor cells is stimulated and/or increased. MVX-ONCO-2 is composed of a cell suspension of irradiated autologous tumor cells and two capsules loaded with allogenic genetically modified cells releasing an immunomodulator, granulocyte-macrophage colony stimulating factor (GM-CSF). MVX-ONCO-2 is an evolution of MVX-ONCO-1, which was approved for clinical investigation under the same category in a phase I and a phase II clinical trials. The objectives of the trial are to investigate the safety, tolerability and signals of efficacy of MVX-ONCO-2 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with advanced metastatic solid tumors with documented tumor progression after at least one line of systemic therapy and for which no further standard therapies are available, feasible or accepted by the patient. Prior exposure to an immune checkpoint inhibitor (ICPI) is allowed. Patient with a localized disease for which no curative therapy is available and a measurable lesion is still amenable for RECIST assessment after biopsy (to manufacture the vaccine) are allowed (example: GBM or sarcoma with local relapse after surgery, chemo-radiation)
* Must be 18 years of age or older at the time of signing the informed consent.
* Must have a primary tumor and/or metastasis amenable for surgery (or tap as indicated).
* Must be willing to undergo a surgical tumor biopsy (or tap as indicated) prior to registration.
* Must have at least 1 additional radiologically measurable lesion of the primary cancer type, evaluable per RECIST 1.1, that will remain untouched by surgical harvest procedure for the assessment of tumor size throughout the study.
* Must have a life expectancy estimate of at least 4 months.
* Must have Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0 to 1.
* Must have no major impairment of liver function: Alanine aminotransferase (ALT) ≤ 2.5 × the upper limit of the normal range (ULN); bilirubin ≤ 1.5 × ULN. Exceptions:

  * Liver metastases: ALT ≤ 5 × ULN; bilirubin ≤ 3 × ULN;
  * Documented diagnosis of Gilbert syndrome: total bilirubin ≤ 3 × ULN.
* Must have no major impairment of renal function: Estimated glomerular filtration rate (eGFR) > 30 mL/min as calculated using the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI).
* Must have no major impairment of bone marrow function (without hematological support within 7 days prior to assessment): Hemoglobin ≥ 9.0 g/dL; complete blood count (CBC) ≥ 2.5 × 109/L; neutrophils ≥ 1.5 × 109/L; platelets ≥ 75 × 109/L.
* Must have no major impairment of coagulation status: International normalized ratio (INR) ≤ 1.5 × ULN (without anticoagulation therapy), prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ ULN.
* May be male or female.

  1. A male participant with a female partner of childbearing potential must agree to remain sexually abstinent or use condoms during the treatment period with MVX-ONCO-2 and for 60 days after the last treatment; and the patient must also refrain from donating sperm during this period.
  2. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  i. Not a woman of childbearing potential (WOCBP). OR ii. A WOCBP who has had a negative pregnancy test within 7 days before the first study treatment and agrees to follow contraceptive guidance during the treatment period and for at least 60 days after the last dose of study treatment.
* Has the ability to understand the concept of a clinical study and be willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures.
* Is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this Protocol.
* Patient or legal representative has signed an ICF prior to any study-specific procedures or treatment.

Exclusion Criteria:

* Has participated in any other investigational study or received an experimental therapeutic procedure considered to interfere with the study in the 4 weeks before Screening.
* Has received any prior cytotoxic biologic or any investigational agent treatment in the 4 weeks (or 5 half-lives, whichever is shorter) before Screening. Chronic treatment with non investigational gonadotropin-releasing hormone analogues or other hormonal or supportive care is permitted.
* Has received prior radiotherapy within 2 weeks of the start of study treatment. Prior irradiation of RECIST 1.1 target lesions is not allowed.

Note: radiotherapy of bone metastases to control pain is allowed.

- Has history of another malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

Note: The time requirement does not apply to patients who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.

* Has known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has known history of positive test for HIV-1 or HIV-2 unless on established anti-retroviral therapy (ART) for at least 4 weeks prior to treatment administration and whose viral load is ≤ 400 copies/mL prior to enrollment.
* Has known history of hepatitis B virus (HBV). Patients who are hepatitis B surface antigen negative and HBV viral deoxyribonucleic acid (DNA) negative may be included in the study. Patients who had HBV but who received an antiviral treatment and show non-detectable viral DNA for 6 months or patients who are seropositive because of HBV vaccine may also be included in the study.
* Has known history of hepatitis C virus (HCV). Patients who had HCV but who received an antiviral treatment and show no detectable HCV viral deoxyribonucleic acid (DNA) for 6 months may be included in the study.
* Has known active or recent cytomegalovirus (CMV) infection.
* Has received vaccine containing live virus within 4 weeks prior to the first dose of study treatment. Inactivated seasonal influenza vaccines are permitted on study without restriction.
* Has a clinically severe auto-immune condition requiring immunosuppressive medication.
* Has a history of transplants.
* Has conditions requiring concurrent use of systemic immunosuppressants or corticosteroids > 30 mg daily of cortisone or equivalents. Topical steroids at or near the injection site should not be allowed.
* Use of other immunosuppressive medications within 14 days of study treatment.
* Has evidence of chronic or concurrent active infection or medical condition that requires intravenous antibacterial, antiviral, or antifungal therapy within 14 days of the first study treatment administration.
* Has other unresolved toxicities related to prior anticancer therapy and/or surgery.

Note: Patient must have stabilized or recovered (Grade 1 or baseline) from all prior therapy related toxic effects of prior therapy or surgical procedure (except alopecia).

* Has uncontrolled or significant cardiovascular disease including, but not limited to, any one of the following:

  * Myocardial infarction ≤ 6 months prior to the first dose;
  * Unstable angina pectoris;
  * Uncontrolled congestive heart failure (New York Heart Association [NYHA] > Class II);
  * Uncontrolled ≥ Grade 3 hypertension (per the CTCAE); and
  * Uncontrolled cardiac arrhythmias.
* Has any known or underlying medical or psychiatric condition, and/or social situations that, in the opinion of the Investigator, would limit participation and compliance with the study requirements.
* Has a history of allergy or hypersensitivity to any of the study treatments or study treatment components.
* Has received transfusions of blood products (including platelets or red blood cells), or the administration of colony-stimulatory factors (including G-CSF and GM-CSF), or recombinant erythropoietin within 4 weeks before the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events and/or serious adverse events | 6 months
  Safety parameters including, but not limited to, adverse events (AEs) and serious adverse events (SAEs) (incidence, causality, severity), changes in laboratory values, and vital signs.

SECONDARY OUTCOMES:
Tumor response | 2 years
  Assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response | 2 years
  Assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression-free survival | Assessed up to 5 years
Overall survival | Assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Fernandez, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No